CLINICAL TRIAL: NCT06749405
Title: Assessment of a Quantra-guided Transfusion Algorithm in Liver Transplantation
Acronym: QUALIVERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/23/0621; 2024-A00944-43 (Other: Agence National de Sécurité du Médicament)
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation; Bleeding; Blood transfusion; Quantra®; Viscoelastic test; Haemorrhagic surgery; Labile blood products; Randomized controlled trial; Coagulation; End-stage liver disease (ESLD)
MeSH Terms: conditions — Hemorrhage; Thrombosis; End Stage Liver Disease

STUDY DESIGN:
Intervention Model Description: * Intervention Group: Patients managed using a transfusion algorithm based on Quantra®
  * Control Group: Patients managed using a conventional transfusion algorithm
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transfusion algorithm based on Quantra® (Experimental): Patients managed using a transfusion algorithm based on Quantra®.
  Interventions: Biological: Transfusion algorithm based on Quantra®
- Conventional transfusion algorithm (Active Comparator): Patients managed using a conventional transfusion algorithm.
  Interventions: Biological: Conventional transfusion algorithm

INTERVENTIONS:
Biological: Transfusion algorithm based on Quantra® — In addition to routine coagulation tests, a Quantra Qstat® analysis will be performed at baseline (before incision), at the end of native liver dissection, and after unclamping of the venous anastomoses. In the event of bleeding, additional Quantra Qstat® analyses may be conducted until bleeding control is achieved.
  Transfusion and administration of blood-derived medications will be guided by the results of the Quantra Qstat® analyses.
  Arms: Transfusion algorithm based on Quantra®
Biological: Conventional transfusion algorithm — Transfusion and blood-derived medications will be guided by the results of routine coagulation tests.
  Arms: Conventional transfusion algorithm

SUMMARY:
Liver transplantation carries a substantial risk of bleeding, making precise haemostasis control essential, although assessing coagulation remains challenging. Quantra, a bedside viscoelastic testing device using sonorheometric methods, offers an innovative approach to guiding haemostatic management during surgery. The study aims to determine whether a Quantra-guided transfusion can reduce transfusion and bleeding during liver transplantation when compared to a conventional transfusion approach.

DETAILED DESCRIPTION:
Liver orthotopic transplantation (LT) represents the best treatment option for patients with end-stage liver disease (ESLD), as well as for various oncological, metabolic, and genetic indications. In the setting of ESLD, particularly when decompensated, LT is associated with a substantial risk of bleeding, making the assessment of coagulation and haemostasis management challenging. ESLD is characterized by a fragile balance between pro- and anti-coagulant factors, where routine coagulation tests are often altered but poorly correlated with the risk of bleeding. Additionally, the presence of portal hypertension with venous collaterals and previous abdominal surgeries significantly increase surgical risk. Many intraoperative events, such as acidosis, hypocalcaemia, consumptive coagulopathy, haemodilution, or post-reperfusion hyperfibrinolysis are also likely to induce or exacerbate bleeding. These factors highlight the challenges anaesthesiologists face when guiding haemostatic management during LT. A transfusion strategy based on routine coagulation tests is widely questioned. These tests provide an imperfect reflection of clot formation in cirrhotic patients, fail to assess haemostasis comprehensively, and do not consider the coagulation-anticoagulation balance. Moreover, the minimum delay in obtaining biological results (typically around 30 to 60 minutes), complicates this therapeutic approach, particularly in bleeding emergencies, when the biological findings no longer fully reflect the clinical situation at the time of receiving the results.

Viscoelastic tests (VETs) offer a better understanding of haemostatic capacity and can guide the transfusion of labile blood products. VETs dynamically evaluate clot formation, encompassing processes from platelet activation to fibrinolysis. As rapid functional assays, they pinpoint the specific disruptions in the coagulation process and assist clinicians to determine the most appropriate haemostatic intervention. Several studies have demonstrated that implementing VET-guided transfusion algorithms in LT can reducethe use of therapeutic plasma and red blood cell concentrates, potentially decreasing perioperative bleeding. Despite these advantages, the routine adoption of VETS in clinical practice faces significant technical challenges, particularly in the management of pre-analytical and analytical phases, as well as in the interpretation of result.

The Quantra® (Stago BioCare) is a next-generation coagulation monitoring device that assesses the viscoelastic properties of clot formation through sonorheometry. By avoiding mechanical contact, it offers an innovative approach with high sensitivity to weak clots, particularly in cases of hypofibrinogenemia or thrombocytopenia. and its use is simplified by ready-to-use cartridges. However, the clinical relevance of a Quantra®-based transfusion algorithm in LT-specifically for transfusion reduction and bleeding management-has yet to be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patient with ESLD undergoing liver transplantation
* Individuals affiliated with or beneficiaries of a social security scheme
* Free and informed written consent obtained in writing from the patient, or where applicable from the trusted person/family member/close relative

Non-inclusion Criteria:

* Multi-organ transplantation
* Congenital haemostasis disorder (such as haemophilia)
* Patient under juridical protection (persons deprived of liberty or under curatorship or guardianship or safeguard of justice)
* Pregnant or breast-feeding woman
* Patient already enrolled in another interventional study with primary or secondary objective of reducing perioperative bleeding or transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-03-08 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Fresh Frozen Plasma (FFP) transfusion during liver transplantation surgery | Conducted during surgery
  Number of FFP transfused intraoperatively during liver transplantation surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume PORTA BONETE, Md, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, France